CLINICAL TRIAL: NCT05027321
Title: Efficacy of Preparation in Self-Hypnosis by Anchoring Versus Conversational Hypnosis, Used Alone or Combined, in Patients Undergoing Breast Macrobiopsies: a Randomized Study
Brief Title: Efficacy of Preparation in Self-Hypnosis by Anchoring Versus Conversational Hypnosis, Used Alone or Combined, in Patients Undergoing Breast Macrobiopsies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HYACOM
Record Dates: First submitted 2021-08-16; First posted 2021-08-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Neoplasm Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): control
- Preparation in Self-Hypnosis by anchoring (Experimental): 1-hour consultation with a hypnopractor just before the examination
  Interventions: Behavioral: Preparation in Self-Hypnosis by anchoring
- Conversational Hypnosis (Experimental): conversational hypnosis support during the examination by a radiology technician and a radiologist specifically trained
  Interventions: Behavioral: Conversational Hypnosis
- Preparation in Self-Hypnosis by anchoring + Conversational Hypnosis (Experimental): 1-hour consultation with a hypnopractor just before the examination and conversational hypnosis support during the examination by a radiology technician and a radiologist specifically trained
  Interventions: Behavioral: Preparation in Self-Hypnosis by anchoring + Conversational Hypnosis

INTERVENTIONS:
Behavioral: Preparation in Self-Hypnosis by anchoring — Preparation in Self-Hypnosis by anchoring just before examination
  Arms: Preparation in Self-Hypnosis by anchoring
Behavioral: Conversational Hypnosis — Conversational Hypnosis during examination
  Arms: Conversational Hypnosis
Behavioral: Preparation in Self-Hypnosis by anchoring + Conversational Hypnosis — Preparation in Self-Hypnosis by anchoring just before examination combied with Conversational Hypnosis during examination
  Arms: Preparation in Self-Hypnosis by anchoring + Conversational Hypnosis

SUMMARY:
The incidence of breast cancer and its mortality are reduced thanks in particular to early detection.

Often performed after a screening test, stereotactic macrobiopsies are used to characterize abnormalities detected on mammography. This anxiety-inducing and painful examination leads to significant physiological and psychological modifications for these women who logically apprehend the realization of this act.

Faced with this observation, investigators wondered what could be done to improve the experience of the patients during this examination.

Investigators were interested in hypnosis because its effectiveness as a complementary practice has been validated by numerous studies with benefits on pain and stress management.

However, today, there are no convincing results confirming which hypnosis method would be the best to manage patients' anxiety and pain during this examination.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or over,
* referred to the medical imaging department of Saint-Joseph hospital for breast macrobiopsy,
* naive of any hypnosis,
* having given free, informed and written consent,
* being affiliated to a social security scheme or beneficiary of such scheme

Exclusion Criteria:

* having a major hearing loss,
* suffering from identified mental or psychotic disorders,
* not understanding the French language,
* having already had hypnosis practices,
* having an ongoing pregnancy,
* being the subject of a safeguard measure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
change in anxiety score | baseline (pre-intervention, during the intervention, immediatly after the intervetion) and at 8 days
  Score (from 20 to 80) measured on the State-Trait Anxiety Inventory for state anxiety (STAI-Y1), how respondent feels right now, at this moment.
  Total scores can be categorized into five levels:
  1. > 65 (very high),
  2. from 56 to 65 (high),
  3. from 46 to 55 (medium),
  4. from 36 to 45 (low),
  5. < 35 (very low). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
change in anxiety score | baseline (pre-intervention, during the intervention, immediatly after the intervetion) and at 8 days
  measured on anxiety visual analog scale from 0 (not at all anxious) to 8 (extremely anxious)
change in pain score | baseline (pre-intervention, during the intervention, immediatly after the intervetion) and at 8 days
  measured on pain visual analog scale from 0 (no pain) to 10 (worst pain)
patient examination experience | baseline (immediately after the intervention)
  measured on satisfaction visual analog scale from 0 (poor experience quality) to 10 (very good experience quality)
staff examination experience | baseline (immediately after the intervention)
  measured on satisfaction visual analog scale from 0 (poor experience quality) to 10 (very good experience quality)
anxiety score | baseline (pre-intervention)
  STAI-Y2 (score from 20 to 80 measured on the STAI for trait anxiety), how respondent generally feel
  Total scores can be categorized into five levels:
  1. > 65 (very high),
  2. from 56 to 65 (high),
  3. from 46 to 55 (medium),
  4. from 36 to 45 (low),
  5. < 35 (very low). Higher scores mean a worse outcome.
Amount of nesthetic administered to the patiet during the procedure | baseline (immediately after the intervention)
  mL
Examination duration | baseline (immediately after the intervention)
  minutes
AE/SAE reporting | baseline (during the intervention, immediatly after the intervetion) and at 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Joseph, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided